CLINICAL TRIAL: NCT01613885
Title: Understanding and Diagnosing Allergic Disease in Twins
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kari Christine Nadeau, MD, PhD, Associate Professor, Stanford University
Other Study IDs: SU-10042011-8546
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Allergies
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, nasal /cheek/throat/skin swab, saliva, urine, stool, sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Twins: Twins that are ages 0 to 80 years, with or without allergy disease.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This study does not involve any intervention other than obtaining blood, nasal/cheek/throat/skin swabs, saliva, sputum, urine, and stool samples, breathing and skin tests.

SUMMARY:
The purpose of this study is to gain better understanding of how the immune system works in twins with and without allergic disease. Healthy volunteers are not specifically targeted. Healthy non-allergic study participants may be found through the course of evaluation for the presence of allergies.

DETAILED DESCRIPTION:
The purpose of this study is to study the genetic control and gain better understanding of how the immune system works in twins with and without allergic disease. Although healthy volunteers are not specifically targeted, they might be identified when non-allergic study participants are found through the course of evaluation for the presence of allergies.

ELIGIBILITY:
Inclusion Criteria:

* Twin participants ages 0 to 80 years who are with or without allergy disease.

Exclusion Criteria:

* Patients with special risks attendant to venipuncture will be excluded.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers are not specifically targeted. Healthy non-allergic study participants may be found through the course of evaluation for the presence of allergies. Women, minorities or children will not be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Comparing immune systems of food allergic twins | 2 years
  Differences in genetic and phenotypic characteristics between twin siblings

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Sean N Parker Center for Allergy and Asthma Research at Stanford, Stanford, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Derived] Bao R, Hesser LA, He Z, Zhou X, Nadeau KC, Nagler CR. Fecal microbiome and metabolome differ in healthy and food-allergic twins. J Clin Invest. 2021 Jan 19;131(2):e141935. doi: 10.1172/JCI141935. PMID 33463536